CLINICAL TRIAL: NCT02755740
Title: Promoting Smoking Cessation for Female Smokers in Hong Kong Through Training Female Youth Smoking Cessation and Reduction Ambassadors (SCRA)
Brief Title: Promoting Smoking Cessation for Female Smokers in Hong Kong Through Training Female Youth SCRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Girl Guide
Record Dates: First submitted 2016-04-17; First posted 2016-04-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Smoking Cessation
Keywords: female
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- receiving age and gender-specific SC advice (Other): After delivering the "AWARD" advice, the trained SCRA will seek consent from and refer adult female smokers (aged over 25 years) to our intensive smoking cessation telephone or face-to-face counselling interventions, which has already counselled 509 female smokers with a quit rate of 29.7% at 6-month and 26.7% at 3-year follow up. Female youth smokers will give consent and be referred to our Youth Quitline (5111 4333), a smoking cessation telephone counselling for young people aged 25 or below which has counselled 1257 smokers with a quit rate of 21.9% at 6 months. If necessary, the female smokers can be referred to other smoking cessation services (e.g., the integrated smoking cessation hotline by the Department of Health (1833-183).
  Interventions: Other: receiving age and gender-specific SC advice

INTERVENTIONS:
Other: receiving age and gender-specific SC advice — After delivering the "AWARD" advice, the trained SCRA will seek consent from and refer adult female smokers (aged over 25 years) to our intensive smoking cessation telephone or face-to-face counselling interventions, which has already counselled 509 female smokers with a quit rate of 29.7% at 6-month and 26.7% at 3-year follow up. Female youth smokers will give consent and be referred to our Youth Quitline (5111 4333), a smoking cessation telephone counselling for young people aged 25 or below which has counselled 1257 smokers with a quit rate of 21.9% at 6 months. If necessary, the female smokers can be referred to other smoking cessation services (e.g., the integrated smoking cessation hotline by the Department of Health (1833-183).

SUMMARY:
This project aims to promote quitting, and reduction for those who do not want to quit, among female smokers through training female youth as smoking cessation and reduction ambassadors (SCRA). The objectives are to:

1. Promote age and gender-specific smoking cessation and reduction to the female population
2. Deliver a smoking cessation and reduction ambassador training workshop to equip and empower female youth with the knowledge on the adverse effects of smoking on female smokers and the skills in smoking cessation and reduction and in raising public awareness of the harmful effects of smoking on female smokers.
3. Have the trained female youth to deliver a brief advice (AWARD) to female smokers to help them to quit or reduce smoking and refer them to the female-specific smoking cessation hotline or the Department of Health Quitline for further assistance if needed.

DETAILED DESCRIPTION:
Phase I: Increase public awareness of the beneficial effects of smoking cessation on female smokers Five thousand leaflets on woman smoking cessation will be distributed to the Girl Guide, the University of Hong Kong and 40 secondary schools. For those who are not ready to join the training, they will be encouraged to help to increase the awareness of the importance of promoting smoking cessation by disseminating the leaflets to others, especially female smokers in the population.

Phase II: Deliver a smoking cessation training curriculum for the female youth recruited through the Hong Kong Girl Guides Association, the University of Hong Kong and 40 secondary schools.

The investigators aim to train 120-150 female youth (with the priority given to the Hong Kong Girl Guides Association) to be SCRA with better understanding on the needs and feelings of female smokers.The investigators will deliver a half-day SCRA training workshop to the female youth. In addition to the leaflets above, the investigators shall publicize the training workshop and recruit participants via bulk emails, newsletters and the homepage of the Hong Kong Girl Guides Association, the University of Hong Kong and 40 secondary schools. The investigators will draw on our experience in conducting smoking cessation training programmes for our existing projects such as Youth Quitline and Quit to Win Contests. In addition, the investigators shall train and empower participants how to deliver a brief smoking cessation advice to female smokers. For those who do not want to quit, they will be advised to reduce smoking as the first step towards quitting. Throughout the training, participants will be taught to deliver the "AWARD" approach: 1) Ask about smoking, 2) Warn the smokers that at least half will be killed by smoking, and the female specific harms due to smoking, 3) Advise to quit (or reduce) as soon as possible, 4) Refer to a cessation clinic or hotline, and 5) Do it again until they quit.7 At the end of the training workshop, participants should be capable of delivering brief smoking cessation and reduction advice to female smokers, and a referral system will be set up so that women who accept more intensive counselling can be referred to our and other more specialised smoking cessation services. Upon completion of the training, a certificate of attendance will be awarded to the participants.

The outcomes of the training will be evaluated before and immediately afterwards, and 3- and 6-month post training. A smoking-, tobacco control-, and smoking cessation and reduction-related knowledge, attitudes and practice (KAP) survey, 15 using a modified version of previous questionnaires which have been used to assess other smoking cessation training workshop,16 will be conducted.

Additionally, there is increasing evidence that the Health Action Process Approach (HAPA) is helpful in explaining the psychological mechanisms in bridging the gap between intention and actual change in health behaviour.17 According to HAPA model, an individual's intention either to engage in a preventive measure or to modify risky behaviour in favour of a healthy practice, action plans and action control help the individual to structure a strategy for maintaining healthy practices and defeating other conflicting ideas.18 Adopting the HAPA model,17 intention, self-efficacy, and planning to provide smoking cessation and reduction advice will also be assessed.

Phase III: Deliver a age and gender-specific smoking cessation advice

The trained female SCRA will be encouraged to deliver "AWARD" to at least 2 female smokers to advise them to reduce and quit smoking. Self-help smoking cessation booklet designed by Hong Kong Council on Smoking and Health, a partner of our smoking cessation research team, will be provided. The trained youth ambassadors can identify and reach the target female smokers in the following ways:

1. from their family members, relatives, friends, peers, schoolmates, or colleagues in workplaces;
2. If the trained youth ambassadors cannot identify and reach target female smokers from (1), the investigators can refer female smokers to them through our other smoking cessation projects, such as Youth Quitline or Quit to Win project with the consensus from the female smokers

ELIGIBILITY:
Inclusion Criteria:

* be able to communicate with Cantonese

Exclusion Criteria:

* taking Psychiatric drugs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The self-reported quit rate | 6-month follow-up
  not smoke for at least 7 days

SECONDARY OUTCOMES:
biochemical-validated quit rate | 6-month follow-up
  measurement of exhaled (CO) and salivary cotinine level
smoking reduction rate | 1-, 3-, and 6-month follow-up
smoking quit attempt | 1-, 3-, and 6-month follow-up
KAP change of SCRA from baseline to 3- and 6-month follow-up | 3- and 6-month follow-up
  Use questionnaires to measure the change of smoking cessation and reduction-related knowledge, attitudes and practice of Smoking Cessation Ambassadors.

CONTACTS AND LOCATIONS:
Overall Officials: William LI, Phd, Principal Investigator — School of Nursing, the University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No